CLINICAL TRIAL: NCT04534075
Title: Dietary Fiber During Radiotherapy and Intestinal Inflammation - a Placebo-controlled Randomized Trial (FIDURA)
Brief Title: Dietary Fiber During Radiotherapy - a Placebo-controlled Randomized Trial
Acronym: FIDURA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: The Swedish Research Council (Other Government); VGregion (Unknown); Sjöbergstiftelsen (Unknown)
Responsible Party: Principal Investigator, Gunnar Steineck, Senior Professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ALFGBG-926 421; 2018-02966 (Other: Swedish Research Council); 2020-01-07-02 (Other: Sjöbergstiftelsen)
Record Dates: First submitted 2020-08-22; First posted 2020-09-01 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Malignant Neoplasm; Malignant Neoplasm of Rectum; Malignant Neoplasm of Anus; Malignant Neoplasm of Urinary Bladder; Malignant Neoplasm of Cervix; Malignant Neoplasm of Ovary; Malignant Neoplasm of Prostate; Malignant Neoplasm of Large Intestine; Malignant Neoplasm of Colon; Gynecologic Cancer
Keywords: Radiotherapy; Irradiation; Radiation therapy; Dietary fiber; Psyllium husk; Placebo-controlled; Double-blind; Randomized; Patient-reported outcomes; ePROMS; Gut-wall inflammation; Late adverse effects; Late effects; Treatment-induced cancer survivorship diseases; Treatment-induced cancer survivorship syndromes; Intestinal health; Bowel health; Urgency; Leakage; Mucus; Flatulence; Blood discharge
MeSH Terms: conditions — Neoplasms; Rectal Neoplasms; Anus Neoplasms; Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Colonic Neoplasms; Flatulence

STUDY DESIGN:
Intervention Model Description: Random allocation of patients and blinding of researchers, patients, healthcare professionals and outcome assessors.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Capsules that look alike, with dietary fiber or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Additional dietary fiber through Psyllium husk (Experimental): The participants are allocated to intake the fifteen capsules per day, for example, five capsules three times per day. Altogether the fifteen capsules contains 5.5 g dietary fiber in psyllium husk.
  Interventions: Biological: Capsules containing either dietary fiber or placebo
- Placebo (no additional dietary fiber) (Placebo Comparator): The participants are allocated to intake the fifteen capsules per day, for example, five capsules three times per day. The capsules contain placebo (maltodextrin) and have a similar look as in the experimental arm.
  Interventions: Biological: Capsules containing either dietary fiber or placebo

INTERVENTIONS:
Biological: Capsules containing either dietary fiber or placebo — The participants are invited to eat 15 capsules per day. The capsules either contain dietary fiber from psyllium husk or placebo.

SUMMARY:
The investigators hypothesize that an increase in dietary fiber intake during radiation therapy may provide better long-term intestinal health for the cancer survivor. If the hypothesis is not correct, the increased intake may only mean an increase in acute side effects. All participants are advised to consume at least 16 g of dietary fiber/day via food. In addition, participants are invited to take capsules that together contain either 5.5 g of dietary fiber from psyllium husk or placebo.

DETAILED DESCRIPTION:
The overall working hypothesis is that intake of dietary fiber during radiotherapy can mitigate or hinder end states or the triggering of long-lasting pathophysiological processes that decreases intestinal health in the cancer survivor. If correct, there is a dose-effect relationship to be documented. Moreover, if correct, different kinds of dietary fibers may have different effects. Mechanisms for the mitigatory effects may be that dietary fiber helps to preserve the two protective mucus layers and hinder gut-wall starvation. Lack of protection, as well as gut-wall starvation, may decrease the gut walls' integrity. That, in turn, may enhance bacterial migration from the lumen into the gut wall, causing unnecessary inflammation. This inflammation may, in turn, lead to a number of different pathophysiological processes, including a chronic self-propagating low-grade inflammation. Clinical experience suggests the intake of dietary fiber during radiotherapy may increase acute intestinal side effects. Our own data suggest a modest, if any, increase by dietary fiber.

Through recipes of tasty meals by price-winning chefs and general advice, the investigators guide the participant to try to consume at least 16 g of dietary fiber per day via food. The guidance takes place through telephone calls, calls via video link, and text on a website or paper material. The participant gets access to a mobile application that measures the daily intake of dietary fiber. Dietary fiber is ingested in 15 capsules with psyllium husk which contains a total of 5.5 g of dietary fiber. The investigators ask the participant to take the capsules two weeks before radiotherapy, during radiotherapy, and to stop four weeks after the end of radiotherapy. Placebo capsules (maltodextrin) are taken in the same way. To document the frequency of acute side effects, and what symptoms they cause, the participant is asked to report patient-reported outcomes once a week via a mobile application. They are also welcome to report side effects to the study office.

One month after the end of radiotherapy, the degree of inflammation is measured via markers in the blood and feces. One year after the end of radiotherapy, intestinal health is measured via patient-reported outcomes. Blood and feces are collected and patient-reported outcomes are reported in questionnaires and a mobile application before, during, and at least one year after the end of radiotherapy. This data will be a source of in-depth analysis. Radiotherapy gives rise to increased intensity of five different syndromes, fecal-leakage syndrome, urgency syndrome, uncontrolled flatulence, excess mucus discharge, and anal blood discharge. Damage of nerves and small vessels, weakening the anal-sphincter function by muscle fibers turning into the connective tissue (fibrosis), may explain some of the intensity of the fecal-leakage syndrome. An ongoing self-propagating low-grade inflammation, small-vessel and nerve damage in the gut wall may be related to urgency. Reasonably the microbiome, and the communication between the microbiome and the gut wall, is related to uncontrolled flatulence and excess mucus discharge. It is not known to what extent telangiectasias on a fibrotic inner gut wall explains anal blood discharge. Ad hoc studies in FIDURA will explore suggested mechanisms.

An interim analysis will be performed for the primary outcome to identify if there is any effect of the intervention, to decide whether to continue or terminate the inclusion of patients in the study. The concentration of c-reactive protein will be analyzed for all included patients who have donated blood to date (May 2023). To ensure that the blinding is not revealed, all analyses (biochemical and statistical) will be made by external personnel not included in the research group. The capsules are marked with X and Y, and the code for which is intervention or placebo will not be revealed even for the external personnel performing the interim analysis.

ELIGIBILITY:
Inclusion Criteria:

* Planned preoperative (neoadjuvant) or curative radiation therapy for a tumor in the pelvic cavity (including all forms of gynecological cancer, colorectal cancer, anal cancer, prostate cancer, and urinary bladder cancer).

Exclusion Criteria:

* Preoperative stoma which, according to the attending physician, prevents participation
* Difficulty swallowing or ileus conditions which, according to the treating physician, prevent participation
* Cognitive dysfunction which, according to the treating physician, prevents participation
* Need for an interpreter to communicate in Swedish

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2024-09-14 (Actual); Study Completion 2024-09-14 (Actual)

PRIMARY OUTCOMES:
Sign of inflammation i blood | One month after the end of radiotherapy
  Concentration of c-reactive protein in plasma or serum
Intensity of the urgency syndrome | One year after the end of radiotherapy
  Patient-reported outcomes through a validated questionnaire. The metric for the intensity of the urgency syndrome weighs the frequency of several symptoms by factor loadings, as described in PubMed ID 28158314. Examples of the previous usage can be seen in PubMed ID 28366105 and PubMed ID 30601820.

SECONDARY OUTCOMES:
Tolerance to additional dietary fiber | During radiotherapy
  Deviation from the recommended intake of 15 capsules per day
Signs of inflammation i blood | One month after the end of radiotherapy
  Concentration of selected markers in blood and feces. The selection of cytokines and chemokines for this outcome is work in progress 26 august 2020 and will be be given as updated information later on. In feces we will primarily use elastase and calprotectin.
Intensity of the fecal-leakage syndrome, uncontrolled flatulence, excess mucus discharge and blood | One year after the end of radiotherapy
  Patient-reported outcomes through a validated questionnaire. The metric for the intensity of the syndromes weighs the frequency of several symptoms by factor loadings, as described in PubMed ID 28158314. Examples of the previous usage can be seen in PubMed ID 28366105 and PubMed ID 30601820.
Acute side-effects | During radiotherapy, primarily during week 3
  Distress from gastrointestinal symptoms as reported through a mobile phone application (ePROMS). Primarily we ask for defecation frequency, stool consistency (Bristol Scale), and frequency of abdominal pain. The participants may also report other side-effects, either by the mobile phone application, video link, or telephone with the study secretariat.

OTHER OUTCOMES:
Composition of microbiota | During, one month and one year after radiotherapy
  Metrics obtained from freshly frozen defecated feces. The investigators plan to use next-generation sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar N Steineck, MD, PhD, Principal Investigator — Göteborg University; Maria Hedelin, PhD, Study Chair — Göteborg University; Cecilia Bull, PhD, Study Chair — Göteborg University
Locations (1):
- Jubileumskliniken, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
As soon as we we have started publishing data we will successively make our data available to other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From the primary publications and five years afterward.
Access Criteria: Through the Swedish National Data Service, a national data repository run by a consortium consisting of nine universities.
URL: https://snd.gu.se/en

REFERENCES:
- [Background] Patel P, Malipatlolla DK, Devarakonda S, Bull C, Rascon A, Nyman M, Stringer A, Tremaroli V, Steineck G, Sjoberg F. Dietary Oat Bran Reduces Systemic Inflammation in Mice Subjected to Pelvic Irradiation. Nutrients. 2020 Jul 22;12(8):2172. doi: 10.3390/nu12082172. PMID 32707913
- [Background] Malipatlolla DK, Patel P, Sjoberg F, Devarakonda S, Kalm M, Angenete E, Lindskog EB, Grander R, Persson L, Stringer A, Wilderang U, Swanpalmer J, Kuhn HG, Steineck G, Bull C. Long-term mucosal injury and repair in a murine model of pelvic radiotherapy. Sci Rep. 2019 Sep 24;9(1):13803. doi: 10.1038/s41598-019-50023-4. PMID 31551503
- [Background] Hedelin M, Skokic V, Wilderang U, Ahlin R, Bull C, Sjoberg F, Dunberger G, Bergmark K, Stringer A, Steineck G. Intake of citrus fruits and vegetables and the intensity of defecation urgency syndrome among gynecological cancer survivors. PLoS One. 2019 Jan 2;14(1):e0208115. doi: 10.1371/journal.pone.0208115. eCollection 2019. PMID 30601820
- [Background] Ahlin R, Sjoberg F, Bull C, Steineck G, Hedelin M. [Differing dietary advice are given to gynaecological and prostate cancer patients receiving radiotherapy in Sweden]. Lakartidningen. 2018 Oct 9;115:FALY. Swedish. PMID 30325475
- [Background] Sjoberg F, Malipatlolla DK, Patel P, Wilderang U, Kalm M, Steineck G, Bull C. Elastase as a potential biomarker for radiation-induced gut wall injury of the distal bowel in an experimental mouse model. Acta Oncol. 2018 Aug;57(8):1025-1030. doi: 10.1080/0284186X.2018.1438652. Epub 2018 Feb 15. PMID 29447028
- [Background] Bull C, Malipatlolla D, Kalm M, Sjoberg F, Alevronta E, Grander R, Sultanian P, Persson L, Bostrom M, Eriksson Y, Swanpalmer J, Wold AE, Blomgren K, Bjork-Eriksson T, Steineck G. A novel mouse model of radiation-induced cancer survivorship diseases of the gut. Am J Physiol Gastrointest Liver Physiol. 2017 Nov 1;313(5):G456-G466. doi: 10.1152/ajpgi.00113.2017. Epub 2017 Jul 20. PMID 28729245
- [Background] Steineck G, Sjoberg F, Skokic V, Bull C, Wilderang U, Alevronta E, Dunberger G, Bergmark K, Jornsten R. Late radiation-induced bowel syndromes, tobacco smoking, age at treatment and time since treatment - gynecological cancer survivors. Acta Oncol. 2017 May;56(5):682-691. doi: 10.1080/0284186X.2017.1307519. Epub 2017 Apr 1. PMID 28366105
- [Background] Steineck G, Skokic V, Sjoberg F, Bull C, Alevronta E, Dunberger G, Bergmark K, Wilderang U, Oh JH, Deasy JO, Jornsten R. Identifying radiation-induced survivorship syndromes affecting bowel health in a cohort of gynecological cancer survivors. PLoS One. 2017 Feb 3;12(2):e0171461. doi: 10.1371/journal.pone.0171461. eCollection 2017. PMID 28158314
- [Background] Steineck G, Schmidt H, Alevronta E, Sjoberg F, Bull CM, Vordermark D. Toward Restored Bowel Health in Rectal Cancer Survivors. Semin Radiat Oncol. 2016 Jul;26(3):236-50. doi: 10.1016/j.semradonc.2016.03.002. Epub 2016 Mar 18. PMID 27238476
- [Background] Lind H, Alevronta E, Steineck G, Waldenstrom AC, Nyberg T, Olsson C, Wilderang U, Dunberger G, Al-Abany M, Avall-Lundqvist E. Defecation into clothing without forewarning and mean radiation dose to bowel and anal-sphincter among gynecological cancer survivors. Acta Oncol. 2016 Nov;55(11):1285-1293. doi: 10.1080/0284186X.2016.1176247. Epub 2016 May 13. PMID 27173757
- [Background] Thor M, Olsson CE, Oh JH, Petersen SE, Alsadius D, Bentzen L, Pettersson N, Muren LP, Waldenstrom AC, Hoyer M, Steineck G, Deasy JO. Relationships between dose to the gastro-intestinal tract and patient-reported symptom domains after radiotherapy for localized prostate cancer. Acta Oncol. 2015;54(9):1326-34. doi: 10.3109/0284186X.2015.1063779. Epub 2015 Sep 4. PMID 26340136
- [Background] Alsadius D, Olsson C, Pettersson N, Tucker SL, Wilderang U, Steineck G. Patient-reported gastrointestinal symptoms among long-term survivors after radiation therapy for prostate cancer. Radiother Oncol. 2014 Aug;112(2):237-43. doi: 10.1016/j.radonc.2014.08.008. Epub 2014 Sep 4. PMID 25201126
- [Derived] Ahlin R, Bergmark K, Bull C, Devarakonda S, Landberg R, Sigvardsson I, Sjoberg F, Skokic V, Steineck G, Hedelin M. A Preparatory Study for a Randomized Controlled Trial of Dietary Fiber Intake During Adult Pelvic Radiotherapy. Front Nutr. 2021 Dec 7;8:756485. doi: 10.3389/fnut.2021.756485. eCollection 2021. PMID 34950688
- See also: The study's website. Researchers who want to be able to log in, please write to Gunnar.Steineck@gu.se. — https://eftercancern.se/fidura/

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT04534075/SAP_000.pdf